CLINICAL TRIAL: NCT03345784
Title: A Phase I Study of the Wee 1 Kinase (Wee 1) Inhibitor AZD1775 in Combination With Radiotherapy and Cisplatin in Cervical, Upper Vaginal and Uterine Cancers (10041848, 10008224, 10008238, 10046888, 10014735)
Brief Title: Testing AZD1775 inC Combination With Radiotherapy and Chemotherapy in Cervical, Upper Vaginal and Uterine Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00038; NCI-2017-00038 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-01765; PHL-087; 10132 (Other: University Health Network Princess Margaret Cancer Center LAO); 10132 (Other: CTEP); UM1CA186644 (NIH); NCT01958658 (obsolete NCT alias)
Record Dates: First submitted 2017-11-16; First posted 2017-11-17 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Cervical Carcinoma; Endometrioid Adenocarcinoma; Malignant Female Reproductive System Neoplasm; Recurrent Cervical Carcinoma; Stage I Uterine Corpus Cancer AJCC v7; Stage I Vaginal Cancer AJCC v6 and v7; Stage IA Uterine Corpus Cancer AJCC v7; Stage IB Cervical Cancer AJCC v6 and v7; Stage IB Uterine Corpus Cancer AJCC v7; Stage IB2 Cervical Cancer AJCC v6 and v7; Stage II Cervical Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7; Stage II Vaginal Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage III Cervical Cancer AJCC v6 and v7; Stage III Uterine Corpus Cancer AJCC v7; Stage III Vaginal Cancer AJCC v6 and v7; Stage IIIA Cervical Cancer AJCC v6 and v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Vaginal Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Endometrioid; Vaginal Neoplasms | interventions — adavosertib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, adavosertib, cisplatin) (Experimental): Patients undergo external beam radiation therapy on days 1-5 and receive adavosertib PO on days 1, 3, and 5 or QD on days 1-5 and cisplatin IV over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.
  Interventions: Drug: Adavosertib; Drug: Cisplatin; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of adavosertib when given together with external beam radiation therapy and cisplatin in treating patients with cervical, vaginal, or uterine cancer. Adavosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. External beam radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving adavosertib, external beam radiation therapy, and cisplatin may work better in treating patients with cervical, vaginal, or uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II dose (RP2D) and safety profile of adavosertib (AZD1775) in combination with radiotherapy and concurrent cisplatin in patients with gynecological cancers.

SECONDARY OBJECTIVES:

I. To determine the acute and late toxicity of AZD1775 when administered to patients with gynecological cancer in combination with standard radiotherapy and concurrent cisplatin.

II. To evaluate the pharmacodynamic effects of AZD1775 when administered in combination with radiotherapy and concurrent cisplatin (in particular, for the 15 patients treated in an expansion cohort at the RP2D).

III. To obtain preliminary information about the progression-free survival, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or clinical progression, of AZD1775 in combination with standard radiotherapy and concurrent cisplatin in women with gynecological cancer.

OUTLINE: This is a dose-escalation study of adavosertib.

Patients undergo external beam radiation therapy on days 1-5 and receive adavosertib orally (PO) on days 1, 3, and 5 or once daily (QD) on days 1-5 and cisplatin intravenously (IV) over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days and then every 4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following biopsy proven gynecological cancer and a decision to treat with radiotherapy and concurrent cisplatin chemotherapy (RT-CT)

  * Newly diagnosed epithelial carcinoma of the cervix, cT1B-3B, N0/1, M0/1

    * Patient may have small volume metastatic disease in para-aortic or supraclavicular lymph nodes or at other metastatic sites as long as, in the best judgment of the treatment team, a radical course of pelvic radiotherapy is warranted to assure local disease control
  * Newly diagnosed epithelial carcinoma of the upper 1/3 vagina, T1-3, N0/1, M0/1

    * Patient may have small volume metastatic disease in para-aortic or supraclavicular lymph nodes or at other metastatic sites as long as, in the best judgment of the treatment team, a radical course of pelvic radiotherapy is warranted to assure local disease control
  * Newly diagnosed endometrioid adenocarcinoma of the uterus, cT1-3, N0/1, M0 unsuitable for primary surgery because of the extent of local disease; these patients are eligible if a prior decision has been made to treat radically with neoadjuvant chemoradiation followed by surgery or further radiotherapy (including brachytherapy) depending on response
  * Central pelvis or sidewall recurrence of epithelial carcinoma of the cervix of endometrioid adenocarcinoma of the uterus after previous surgery without previous pelvic radiotherapy
* Patients must be planned to receive whole pelvic radiotherapy to a total dose of 45 Gy or greater
* Patients must be able to receive weekly cisplatin
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL

  * Blood transfusions are allowed at any time during the screening, treatment or follow-up period, according to the center recommendations
* Prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR) =< 1.5 upper limit of normal (ULN)
* Total bilirubin: serum bilirubin within normal limits (WNL) or =< 1.5 x ULN in patients with liver metastases; or total bilirubin =< 3.0 x ULN with direct bilirubin WNL in patients with documented Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN) or =< 5 x ULN if known hepatic metastases
* Creatinine clearance (CrCl) >= 60 mL/min as calculated by the Cockcroft-Gault method
* Patients must be able to swallow whole capsules
* The effects of AZD1775 on the developing human fetus are unknown; the preclinical chromosomal aberrations assays have shown potential to induce chromosomal aberrations; in addition, cisplatin and radiotherapy are known to be teratogenic; for this reason, women of child-bearing potential must agree to use two birth control methods (two barrier methods or a barrier method plus a hormonal method) or abstinence prior to study entry, for the duration of study participation prior to study entry, for the duration of study participation, and for 4 months after coming off study; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Females with child-bearing potential must have had a negative serum pregnancy test result =< 28 days prior to the first dose of study treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received any radiotherapy or chemotherapy for their current gynecological cancer
* Patients who received prior pelvic radiotherapy for any indication
* Patients who have a mean resting correct corrected QT (QTc) interval using the Fridericia formula (QTcF) > 470 msec (as calculated per institutional standards) obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart at study entry, or congenital long QT syndrome; AZD1775 should not be given to patients who have a history of Torsades de pointes unless all risk factors contributed to Torsades have been corrected; AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction
* Patients requiring para-aortic radiotherapy
* Patients who are receiving any other investigational agents or anticancer therapy concurrently or within 4 weeks (i.e. 28 days)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD1775 or cisplatin
* Uncontrolled intercurrent illness including, but not limited to, myocardial infarction within 6 months, congestive heart failure, symptomatic congestive heart failure, unstable angina pectoris, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, active liver disease or cerebrovascular disease with previous stroke, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD1775 and chemoradiation are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD1775 and cisplatin, breastfeeding must be discontinued if the mother is treated with AZD1775 and cisplatin; these potential risks may also apply to other agents used in this study
* Patients with another uncontrolled malignancy; patients with a previous malignancy, treated curatively and without evidence of disease relapse are eligible
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD1775; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* History of active clinically significant bleeding
* History of bowel obstruction or malabsorption syndromes (within the last 3 months) which might limit the absorption of the study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (8):
- United States (6):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 5 academic centers in the United States (four sites) and Canada (one site). It enrolled participants from May 2018 to July 2020.
Groups:
- Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1: Patients undergo external beam radiation therapy (45-50Gy) on days 1-5, receive 100mg AZD1775 PO on days 1, 3, and 5, and receive 40 mg/m2 cisplatin IV over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.
- Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1: Patients undergo external beam radiation therapy (45-50Gy) on days 1-5, receive 100mg AZD1775 PO on days 3 and 5, and receive 40 mg/m2 cisplatin IV over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
Started | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 48 [43 to 78] | 53 [35 to 63] | 50.5 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 1 | 3
  United States | 3 | 4 | 7
ECOG Performance Status [Count of Participants; unit: Participants] — 0-Normal activity. Fully active, able to carry on all pre-disease performance w/o restriction. 1-Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory & able to carry out work of a light/sedentary nature. 2-In bed <50% of the time. Ambulatory & capable of all self-care, but unable to carry out any work activities. Up & about >50% of waking hours. 3-In bed >50% of the time. Capable of only limited self-care, confined to bed/chair >50% of waking hours. 4-100% bedridden. Completely disabled. Cannot carry on any self-care. Totally confined to bed /chair. 5-Dead.
  Participants
    0 | 1 | 4 | 5
    1 | 4 | 1 | 5
Primary Site [Count of Participants; unit: Participants]
  Cervical | 4 | 5 | 9
  Uterine | 1 | 0 | 1
Prior Therapy [Count of Participants; unit: Participants]
  Surgery | 5 | 5 | 10
  Radiation | 0 | 0 | 0
FIGO Stage [Count of Participants; unit: Participants] — Describes the extent of cancer in the body. The extent increases with stage.
  Participants
    IA | 1 | 0 | 1
    IB | 1 | 1 | 2
    IIA | 1 | 1 | 2
    IIB | 1 | 1 | 2
    IIIB | 1 | 2 | 3
Grade [Count of Participants; unit: Participants] — The grade of a cancer tells you how much the cancer cells look like normal cells. Lower grades look most like normal cells while higher grades look more abnormal.
  Participants
    1 - Low grade (well differentiated) | 2 | 0 | 2
    2 - Intermediate grade (moderately differentiated) | 1 | 3 | 4
    3 - High grade (poorly differentiated) | 1 | 2 | 3
    Unknown | 1 | 0 | 1
Histology [Count of Participants; unit: Participants]
  Cervical squamous-cell carcinoma | 3 | 5 | 8
  Cervical adenocarcinoma | 1 | 0 | 1
  Uterine endometrioid adenocarcinoma | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose Defined as the Dose Level With < 1/6 Patients With Dose Limiting Toxicities
Description: To determine the recommended phase II dose (RP2D) and safety profile of AZD1775 in combination with radiotherapy and concurrent cisplatin in patients with gynecological cancers.
Time Frame: Up to week 5
Population: Participants that were evaluable for response.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1: Patients undergo external beam radiation therapy on days 1-5, receive AZD1775 PO on days 1, 3, and 5, and receive cisplatin IV over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.
- Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1: Patients undergo external beam radiation therapy on days 1-5, receive AZD1775 PO on days 3 and 5, and receive cisplatin IV over 1 hour on day 1 or 3. Cycles repeat each week for up to 5 weeks in the absence of disease progression of unacceptable toxicity.
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
Number analyzed (Participants) | 3 | 4
Participants | NA — Could not be determined due to early study closure (due to clinically significant toxicity, slow accrual and significant adverse events also reported with the combination of AZD1775 and chemoradiation in other studies) | NA — Could not be determined due to early study closure (due to clinically significant toxicity, slow accrual and significant adverse events also reported with the combination of AZD1775 and chemoradiation in other studies)

2. Secondary Outcome: Frequency and Severity of AZD1775 Toxicity Events in Patients With Gynecological Cancer in Combination With Standard RT and Concurrent Cisplatin
Description: To determine the acute and late toxicity of AZD1775 when administered to patients with gynecological cancer in combination with standard radiotherapy and concurrent cisplatin. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a subanalysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.
Time Frame: Up to 2 years
Measure: Number; unit: events
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
Number analyzed (Participants) | 4 | 5
events
  All Grade 1-2 Toxicities | 46 | 53
  Related Grade 1-2 Toxicities | 37 | 36
  All Grade 3-4 Toxicities | 8 | 3
  Related Grade 3-4 Toxicities | 8 | 3

3. Secondary Outcome: Pharmacodynamic Effects of AZD1775 in Combination With RT and Concurrent Cisplatin
Description: To evaluate the pharmacodynamic effects of AZD1775 drugs when administered in combination with radiotherapy and concurrent cisplatin. Pharmacodynamic biomarkers will include: pCDC2, Ki67, γH2AX, pH3, and CC3. Associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.
Time Frame: Up to 2 years
Population: Not analyzed as samples were not collected, therefore no data are available.
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-free Survival
Description: To obtain preliminary information about the progression-free survival of AZD1775 in combination with radiotherapy and concurrent cisplatin in women with locally advanced gynecological cancer. Progression is defined a clinical or radiological using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
Number analyzed (Participants) | 3 | 4
Participants
  4 Months Post Treatment: Alive and progression-free post-treatment | 3 | 4
  4 Months Post Treatment: Lost to Follow-Up | 0 | 0
  2 Years Post Treatment: Alive and progression-free post-treatment | 3 | 3
  2 Years Post Treatment: Lost to Follow-Up | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Description: Through regular investigator assessment, regular laboratory testing, etc. Frequency and severity of adverse events were tabulated using counts and proportions.
Arm/Group | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 (N=4) | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1 (N=5)
Grade 3 Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Grade 3 Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiation Therapy, AZD1775 3 Days/Week, Cisplatin) Dose Level 1 (N=4) | Treatment (Radiation Therapy, AZD1775 2 Days/Week, Cisplatin) Dose Level -1 (N=5)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 4 (4)
Fatigue (General disorders) | 3 (3) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Investigations) | 3 (6) | 0 (0) — Platelet count decreased
Anemia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Neutropenia (Investigations) | 1 (2) | 1 (2) — Neutrophil count decreased
Lymphopenia (Investigations) | 1 (2) | 2 (3) — Lymphocyte count decreased
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dermatitis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blister Base Scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Paranoia thoughts (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoid thoughts (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation of our study is the small number of patients enrolled due to premature closure; yet the study showed the limiting toxicities of this triplet combination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03345784/Prot_SAP_000.pdf